CLINICAL TRIAL: NCT06618313
Title: Open-label, Single-arm，Exploratory Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of JCXH-213 in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: One Trial to Evaluate the Safety, Tolerability and Efficacy of JCXH-213 in Patients With r/r B-NHL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Kai Hu, Chief physician, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JCXH-213-001
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: B-Cell Non-Hodgkin Lymphoma-Recurrent; B-Cell Non-Hodgkin Lymphoma-Refractory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JCXH-213 experimental group (Experimental): 4 dose groups will be set in this part, following the dose escalation pattern (accelerated titration combined with a "3 + 3").
  Interventions: Drug: JCXH-213,an mRNA-LNP based in vivo CAR therapy

INTERVENTIONS:
Drug: JCXH-213,an mRNA-LNP based in vivo CAR therapy — JCXH-213 infusion

SUMMARY:
Evaluate the Safety and Efficacy of JCXH-213 in Patients with Relapsed/Refractory B-cell non-Hodgkin Lymphoma

DETAILED DESCRIPTION:
Patient will receive study treatment in the treatment observation period. After the end of the treatment observation period, patients will be allowed to continue to receive treatment if there is no major safety problems and the investigator judges that the patient may continue to benefit.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histopathologically confirmed CD19-positive B-cell Hodgkin lymphoma according to WHO 2022 criteria, including but not limited to pathologically confirmed (1) diffuse large B-cell lymphoma, not otherwise specified (DLBCL, NOS); (2) follicular lymphoma (FL); (3)histologically transformed into diffuse large B-cell lymphoma; (4) primary mediastinal large B-cell lymphoma (PMBCL); (5) High-grade B-cell lymphoma (HGBCL) etc.
* ECOG performance status 0 to 1.
* Existing measurable lesions (Lugano 2014 criteria, as detailed in Appendix 2), meeting one of the following conditions: 1) nodal lesions with a long axis length exceeding 15 mm (short axis length is measurable); 2) extra-nodal lesions with both long axis and short axis lengths exceeding 10 mm.

Exclusion Criteria:

* Patients with other malignant tumors within 5 years before screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local radical prostatectomy, radical ductal carcinoma in situ, and radical thyroidectomy.
* B-cell non-Hodgkin lymphoma with active primary or secondary central nervous system involvement.
* Life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT). | The DLT observation period is 21 days after first infusion of JCXH-213.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Hu, Chief Physician, Principal Investigator — Beijing GoBroad Hospital
Locations (1):
- Department of Lymphoma and Myeloma, Yuhengnan Road, Changping District, Beijing, Beijing, China